CLINICAL TRIAL: NCT04974931
Title: Application of PREVENA (Surgical Incision Protection System) in Reducing Surgical Site Complications Following Reversal of Ileostomy or Colostomy: A Randomized Controlled Trial (PRIC Trial)
Brief Title: Application of PREVENA in Reducing Surgical Site Complications Following Reversal of Ileostomy or Colostomy
Acronym: PRIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Michael Kelly, Consultant Colorectal Surgeon, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: St James Hospital
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Stoma Site Infection; Ileostomy - Stoma; Colostomy Stoma

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, multi-center superiority trial with 2 parallel groups and primary endpoint of surgical site infection at day 7 (after 7-day use of PREVENA) and day 30.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients applied with PREVENA system (Active Comparator): This arm relates to the group of participants applied with PREVANA system post reversal of colostomy/ileostomy.
  Interventions: Device: PREVENA Incision Management System
- Patients applied with conventional dressings (No Intervention): This arm relates to the group of participants applied with conventional dressings post reversal of colostomy/ileostomy

INTERVENTIONS:
Device: PREVENA Incision Management System — Eligible participants, i.e. participants meeting inclusive criteria, will be randomised in equal proportions and divided into two arms. The PREVENA dressings will be applied to the
  Other Names: PREVENA Negative Pressure System
  Arms: Patients applied with PREVENA system

SUMMARY:
Surgical site infections (SSI) remain one of the most common complications associated with reversal of ileostomy and colostomy. In addition to having detrimental impacts on the patient's post-operative course, they also pose significant financial ramifications.

There have been comparative studies in the use of negative pressure wound therapy in reducing surgical site infections.

PREVENA Incision Management System is a type of disposable, customizable and powered negative pressure system designed to help manage and protect surgical incisions and their surrounding environment. It is now commonly used as a surgical wound dressings in the setting of vascular surgeries, post-cesarean infections and colorectal resections.

Our study is designed as a randomised controlled trial to examine if PREVERA therapy as a NPWT is more superior than conventional dressings in reducing the rate of surgical site infections.

DETAILED DESCRIPTION:
Background:

Surgical site infections (SSI) remain one of the most common complications associated with reversal of ileostomy. In addition to having detrimental impacts on the patient's post-operative course, they also pose significant financial ramifications.

The use of Negative Pressure Wound Therapy (NPWT) is one strategy that has been extensively studied in reducing the rate of surgical site infections.

PREVENA Therapy is a form of Incisional Negative Pressure Wound Therapy (INPWT) that has been widely used in the management of closed surgical incisions. They are delivered as prophylactic measures in preventing surgical complications such as surgical site infections.

Trial Design:

This study is designed as a randomized, controlled, open-label, multi-center superiority trial with 2 parallel groups and primary endpoint of surgical site infection at day 7 (after 7-day use of PREVENA) and day 30.

Study Setting The trial will be conducted at two different hospitals located in Dublin, Ireland: St James Hospital - Ireland's largest acute academic teaching hospital (Academic Partner - Trinity College Dublin); Tallaght University Hospital - (Academic Partner - Trinity College Dublin)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old
* Patients undergoing elective reversal of ileostomy/colostomy
* Patients who agree to consent to inclusion and follow-up protocol

Exclusion Criteria:

* Patients who do not fulfil study protocol
* Dressings being removed outside defined time periods
* Patients who do not attend for regular outpatient follow up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
To measure surgical site infection incidence on outpatient follow up post reversal ileostomy/colostomy | Four to Six weeks
  The investigators will be assessing and measuring the incidence of surgical site incidence on follow up appointments

SECONDARY OUTCOMES:
To measure surgical site infection incidence on day 5 post reversal ileostomy/colostomy (or earlier, if deemed fit for discharge prior to day 5) | Five days post reversal ileostomy/colostomy
  The investigators will be assessing and measuring the incidence of surgical site incidence on day 5 post reversal ileostomy/colostomy
To measure the time to wound healing | One to Four weeks
  The investigators will be assessing and measuring the time to wound healing based on the duration and last appointment date of home visits by public healthcare nurses involving wound care management

CONTACTS AND LOCATIONS:
Locations (1):
- St James's Hospital, Dublin, Ireland